CLINICAL TRIAL: NCT02966873
Title: A Randomized Controlled Trial of N-Acetylcysteine for Alcohol Use Disorder and Comorbid Post Traumatic Stress Disorder
Brief Title: Clinical Trial for Alcohol Use Disorder and Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elizabeth Santa Ana, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00056889; 1R01AA025086 (NIH)
Record Dates: First submitted 2016-11-04; First posted 2016-11-17 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Post Traumatic Stress Disorder (PTSD); Addiction; Alcohol Abuse
Keywords: Post Traumatic Stress Disorder (PTSD); Addiction; Alcohol Use Disorder; Cognitive Behavioral Therapy; N-acetylcysteine (NAC)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Behavior, Addictive; Alcoholism | interventions — Acetylcysteine; Therapeutics; Cognitive Behavioral Therapy; X-Rays; Proton Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine (NAC) Treatment Group (Experimental): Participant will receive 12 weeks of Active Treatment NAC (2400 mg) daily, as well as weekly cognitive-behavioral therapy, medication management, and Adverse Event (AE) monitoring.
  Participant will receive one week of study medication at a time from the study physician or the study coordinator. The study medication provided in blister packs in the form of 600 mg tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Interventions: Drug: N-Acetylcysteine (NAC) Treatment; Behavioral: Cognitive Behavioral Therapy (CBT); Other: Functional magnetic resonance imaging (fMRI); Other: Proton magnetic resonance spectroscopy (MRS) Imaging
- Placebo Group (Placebo Comparator): Participant will receive 12 weeks of inactive placebo comparator daily, as well as weekly cognitive-behavioral therapy, medication management, and Adverse Event (AE) monitoring.
  Participant will receive one week of study medication (placebo) at a time from the study physician or the study coordinator. The study medication (placebo) provided in blister packs in the form of 600 mg tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Drug: Inactive Placebo Oral Capsule; Other: Functional magnetic resonance imaging (fMRI); Other: Proton magnetic resonance spectroscopy (MRS) Imaging

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) Treatment — Participant will receive 12 weeks of Active Treatment NAC (2400 mg) daily. The study medication will be provided in blister packs in the form of 600 mg tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Arms: N-Acetylcysteine (NAC) Treatment Group
Behavioral: Cognitive Behavioral Therapy (CBT) — Participant will receive 12 weeks of weekly cognitive-behavioral therapy, medication management, and AE monitoring.
Drug: Inactive Placebo Oral Capsule — Participant will receive 12 weeks of inactive placebo. The study medication will be provided in blister packs in the form of 600 mg tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Arms: Placebo Group
Other: Functional magnetic resonance imaging (fMRI) — Participants will be given the option to complete Functional magnetic resonance imaging (fMRI) at two timepoints (pre-treatment and end of treatment).
  Other Names: Imaging
Other: Proton magnetic resonance spectroscopy (MRS) Imaging — Participants will be given the option to complete magnetic resonance spectroscopy (MRS) at two timepoints (pre-treatment and end of treatment).

SUMMARY:
This is a randomized controlled Phase II clinical trial designed to evaluate the effects of N-acetylcysteine (NAC) in reducing Alcohol Use Disorder (AUD) severity and Post Traumatic Stress Disorder (PTSD) symptomatology among individuals with current AUD and PTSD.

DETAILED DESCRIPTION:
The primary objective of the proposed Phase II study is to evaluate the effects of N-acetylcysteine (NAC), in reducing (1) Alcohol Use Disorder (AUD) severity and (2) Post Traumatic Stress Disorder (PTSD) symptomatology among individuals (N=200) with current AUD and PTSD. We will also use functional magnetic resonance imaging (fMRI) and proton magnetic resonance spectroscopy (MRS) to investigate the neural circuitry and neurochemistry underlying comorbid AUD/PTSD and prognostic indicators of positive treatment response. Secondary objectives are to evaluate the effects of NAC on impairment in associated areas of functioning (e.g., depression, anxiety, sleep, risky behaviors). In order to accomplish this we will (1) employ an intent-to-treat, double-blind, placebo-controlled randomized controlled trial that will consist of 12 weeks of treatment with NAC (2400 mg per day) or placebo medication; (2) examine standardized, repeated dependent measures of clinical outcomes at baseline, week 6, week 12, and 3-, 6-, and 12-month follow-up; and (3) employ advanced neuroimaging methodologies, a laboratory cue paradigm, and collect biologic measures of alcohol consumption. All participants will also undergo weekly individual cognitive behavior therapy sessions (CBT).The following specific aims are proposed:

Specific Aim 1: To determine the efficacy of N-acetylcysteine (NAC), as compared to placebo, in reducing alcohol use severity (i.e., total standard drinks, percent days drinking, abstinence rates) and craving.

Specific Aim 2: To determine the efficacy of N-acetylcysteine (NAC), as compared to placebo, in reducing self-report and clinician-rated PTSD symptomatology.

Specific Aim 3: To use multimodal neuroimaging techniques to investigate the pathophysiology underlying AUD and comorbid PTSD, and prognostic indicators of treatment outcome.

The proposed study will answer critical questions regarding the potential of NAC as an effective pharmacotherapy for AUD and comorbid PTSD, and elucidate possible mechanisms underlying improved outcomes. This study has the particular advantage of building directly on positive preliminary findings by (1) further testing NAC in the treatment of individuals with co-occurring AUD/PTSD using a double-blind, placebo-controlled randomized design; (2) measuring functioning in related areas, such as depression and risky behaviors; (3) employing innovative measurements including neuroimaging and laboratory cue paradigms; and (4) employing a multidisciplinary team of experts who have successfully collaborated in the past and are uniquely qualified to implement this type of investigation. This project is directly responsive to the mission of the National Institute of Alcohol and Alcoholism (NIAAA) and the new AUD/PTSD initiative in that it seeks to evaluate a promising therapeutic agent for the treatment of AUD/PTSD and identify neurobiological mechanisms common to AUD/PTSD as potential treatment targets. The findings from this study have the potential to significantly improve the standard of patient care, advance the comorbidity science in this area, and decrease public health expenditures associated with AUD and comorbid PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; any race or ethnicity; age 18 to 70 years old.
2. Subjects must be able to comprehend English.
3. Meet DSM-5 criteria for current alcohol use disorder (AUD).
4. Meet DSM-5 criteria for current PTSD or subthreshold PTSD. Subjects may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or other anxiety disorders (panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder). The inclusion of subjects with affective and other anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with AUD and PTSD (Brady et al., 2000; Kessler et al., 2005). Subjects may meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for another substance use disorder as long as AUD is the primary substance of choice.
5. Subjects taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before treatment initiation. This is because initiation or change of medications during the course of the trial may interfere with interpretation of results.
6. Must consent to random assignment to N-acetylcysteine (NAC) or placebo.
7. Must consent to complete all treatment and follow-up visits.

Exclusion Criteria:

1. Subjects meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, as the study protocol may be therapeutically insufficient.
2. Subjects with a current eating disorder (bulimia, anorexia nervosa) or with dissociative identity disorder, as they are likely to require specific time-intensive psychotherapy.
3. Subjects experiencing significant withdrawal symptoms, as evidence by a score of 10 or above on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA). These subjects will be referred for clinical detoxification and may be re-assessed for study eligibility after medically supervised detoxification has been completed.
4. Individuals considered an immediate suicide risk or who are likely to require hospitalization during the course of the study for suicidality.

   Women who are pregnant, nursing or not practicing an effective form of birth control.
5. Evidence of liver failure; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 3 times the upper limit of normal; asthma or any clinically significant medical condition that in the opinion of the investigator would adversely affect safety or study participation.
6. Use of carbamazepine, phenytoin, nitrous oxide, methotrexate, 6 azauridine triacetate, or nitroglycerin within the last 14 days or any other medication felt to have a hazardous interaction if taken with NAC.
7. History of childhood or adult seizures of any cause.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudie Back, PhD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - The Charleston Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Back SE, Gray K, Jarnecke AM, Saraiya TC, Santa Ana EJ, Killeen T, Joseph JE, Prisciandaro JJ, Brown DG, Nietert PJ, Stecker T, Rothbaum A, Jones JL, Flanagan JC, Brady KT. N-Acetylcysteine for the Treatment of Co-Occurring Posttraumatic Stress Disorder and Alcohol Use Disorder: A Double-Blind, Randomized Controlled Trial. J Clin Psychiatry. 2025 Aug 27;86(4):25m15803. doi: 10.4088/JCP.25m15803. PMID 40875537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this project was ongoing from June 2016 through June 2021. Prior to the Coronavirus pandemic, recruitment efforts were focused in Charleston, South Carolina (clinics, online, community). In 2020, the study team shifted to a full remote approach and opened recruitment across the continental United States.
Pre-assignment Details: Participants were stratified by alcohol use disorder severity and posttraumatic stress disorder severity. Stratified random block randomization was used to balance the randomization assignment with respect to these strata. The purpose of stratification is to distribute these potential prognostic factors equally across treatment groups.
Groups:
- N-Acetylcysteine (NAC) Treatment Group: Participant will receive 12 weeks of Active Treatment N-Acetylcysteine (NAC) (2400 milligrams [mg]) daily, as well as weekly cognitive-behavioral therapy, medication management, and Adverse Event (AE) monitoring.
  The study medication provided in blister packs in the form of 600 mg tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Cognitive Behavioral Therapy (CBT): All participant will receive 12 weeks of weekly cognitive-behavioral therapy, medication management, and AE monitoring.
- Placebo Group: Participants receive 12 weeks of inactive placebo comparator daily, as well as weekly cognitive-behavioral therapy, medication management, and Adverse Event (AE) monitoring.
  The study medication (placebo) provided in blister packs in the form of 600 milligrams [mg] tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Cognitive Behavioral Therapy (CBT): All participant will receive 12 weeks of weekly cognitive-behavioral therapy, medication management, and AE monitoring.
Period: Overall Study
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Started | 93 | 89
Completed | 77 (N=77 represents 77 participants who provided at least one data point at week 12.) | 74 (N=74 represents 74 participants who provided at least one data point at week 12.)
Not Completed | 16 | 15
Not completed — Lost to Follow-up | 16 | 15

BASELINE CHARACTERISTICS:
Groups:
- N-Acetylcysteine (NAC) Treatment Group: Participant will receive 12 weeks of Active Treatment NAC (2400 milligrams [mg]) daily, as well as weekly cognitive-behavioral therapy, medication management, and Adverse Event (AE) monitoring.
  The study medication provided in blister packs in the form of 600 mg tablets. Each participant will be asked to take two (2) 600 mg tablets in the morning and two (2) 600 mg tablets in the evening.
  Cognitive Behavioral Therapy (CBT): All participant will receive 12 weeks of weekly cognitive-behavioral therapy, medication management, and AE monitoring.
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 93 | 89 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (13.2) | 39.7 (12.4) | 40.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 36 | 33 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 18 | 32
  White | 72 | 66 | 138
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity, % Hispanic | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use Severity
Description: Change in Alcohol Use Severity as measured by standard drinks per day using the Time Line Follow Back (TLFB) to measure alcohol consumption.
  Fewer standard drinks per day represent better outcomes. Greater change in standard drinks per day represents better outcomes.
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: standard drinks per day
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Number analyzed (Participants) | 75 | 73
standard drinks per day | -3.406 (3.738) | -3.934 (.825)

2. Primary Outcome: Change in Alcohol Craving - Obsessive Subscale
Description: Change in Alcohol Craving as measured by the Obsessive Compulsive Drinking Scale (OCDS) to measure the obsessive subscale of alcohol craving.
  The OCDS is a 14-item questionnaire that measures alcohol use and attempts to control drinking. Obsessive subscale includes items 1-6.
  Each item is scored on a scale from 0 to 4. Scores range from 0 to 28, with lower scores representing better outcomes.
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Number analyzed (Participants) | 77 | 73
units on a scale | -2.597 (4.314) | -2.521 (3.738)

3. Primary Outcome: Change in Post Traumatic Stress Disorder Symptom Severity - Clinician Rated
Description: Change in Post Traumatic Stress Disorder symptom severity as measured by Clinician Administered PTSD Scale (CAPS-5) for clinician-rated posttraumatic stress symptoms.
  The CAPS-5 is a 30-item structured interview. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 PTSD symptoms, each with severity scores ranging from 0-4. The overall total severity score for CAPS-5 ranges from 0-80, with lower scores representing better outcomes (less severe PTSD).
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Number analyzed (Participants) | 74 | 73
units on a scale | -11.838 (9.834) | -13.863 (10.87)

4. Primary Outcome: Change in Post Traumatic Stress Disorder Symptom Severity - Self Report
Description: Change in Post Traumatic Stress Disorder (PTSD) symptom severity as measured by the Posttraumatic Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-5](PCL-5) for self-reported symptoms.
  The PCL-5 is a 20-item self-report measure that assesses the 20 symptoms of PTSD. The rating scale is 0-4 for each symptom/item, and overall scores range from 0-80, with lower scores representing better outcomes (less severe PTSD).
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Number analyzed (Participants) | 78 | 74
units on a scale | -15.997 (18.907) | -18.129 (18.37)

5. Primary Outcome: Change in Alcohol Craving - Compulsive Subscale
Description: Change in Alcohol Craving as measured by the Obsessive Compulsive Drinking Scale (OCDS) to measure the compulsive subscale of alcohol craving.
  The OCDS is a 14-item questionnaire that measures alcohol use and attempts to control drinking. Compulsive subscale includes items 7-14.
  Each item is scored on a scale from 0 to 4. Scores range from 0 to 32, with lower scores representing better outcomes.
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Number analyzed (Participants) | 77 | 74
units on a scale | -4.584 (3.971) | -4.905 (4.266)

6. Primary Outcome: Change in Alcohol Use Severity - Percent Days Abstinent
Description: Change in Alcohol Use Severity as measured by the percent days abstinent using the Time Line Follow Back (TLFB) to measure alcohol consumption.
  Greater percentage of days of abstinence represents better outcomes. Greater change in Percent Days Abstinent represents better outcomes.
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: percentage of days abstinent for alcohol
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
Number analyzed (Participants) | 75 | 73
percentage of days abstinent for alcohol | 35.6 (35.2) | 31.7 (34.9)

ADVERSE EVENTS:
Time Frame: Approximately 1 year and 3 months (from start of baseline appointment through 12 week treatment phase and 1 year follow up)
Arm/Group | N-Acetylcysteine (NAC) Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/93 | 1/89
Serious Adverse Events (participants affected / at risk) | 5/93 | 3/89
Other Adverse Events (participants affected / at risk) | 39/93 | 39/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (NAC) Treatment Group (N=93) | Placebo Group (N=89)
Injury/Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Hospitalization from injury/accident.
Ectopic Pregnancy & Ruptured Fallopian Tube (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Surgical procedure to repair ruptured fallopian tube (complication from ectopic pregnancy). Participant was hospitalized.
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Suicidal Ideation - Hospitalization
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Pneumonia - hospitalized
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pancreatitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (NAC) Treatment Group (N=93) | Placebo Group (N=89)
Anxiety (Nervous system disorders) | 2 (4) | 7 (11) — Anxiety Anxiety or Panic Attack Anxiety, worsening
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (5) — Constipation
Gastrointestinal Discomfort (Gastrointestinal disorders) | 21 (23) | 9 (11) — Gastrointestinal Discomfort, non-specified
Headache/Migraine (Nervous system disorders) | 4 (4) | 13 (14) — Headache (including worsening) Migraine(including worsening)
Injury (Injury, poisoning and procedural complications) | 9 (12) | 8 (9) — injury: abscess on hand wound post surgery Injury: back injury from work injury: broken toe (pinky, left foot) Injury: broken tooth injury: infection in hand post-surgery injury: knee injury injury: sprained ankle
Muscle or Joint Pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 10 (16) — Muscle or Joint Pain (neck, back, wrist, rib, side, led)
Nausea (Gastrointestinal disorders) | 9 (9) | 5 (6)
Sinusitis (Infections and infestations) | 3 (3) | 6 (9) — Sinusitis
Viral Upper Respiratory Tract Infections (Cold) (Infections and infestations) | 15 (17) | 14 (17) — Viral Upper Respiratory Tract Infections (Cold)
Flatulence (Gastrointestinal disorders) | 5 (5) | 2 (2) — Flatulence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT02966873/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT02966873/ICF_002.pdf